CLINICAL TRIAL: NCT01238367
Title: Multi-centre, Open-label, Non-randomised Single Dose Trial Investigating the Pharmacokinetics of N8 in Japanese Subjects With Haemophilia A
Brief Title: A Single Dose Trial of Recombinant Factor VIII (N8) in Japanese Subjects With Haemophilia A: An Extension to Trial NN7008-3543
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-3600; U1111-1117-1286 (Other: WHO); JapicCTI-101346 (Other: JAPIC)
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- recombinant factor VIII (N8) (Experimental)
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — Subjects will receive recombinant factor VIII (N8) at a dose of 50 +/- 5 IU/kg body weight. Intravenous administration as a single bolus injection.
  Other Names: N8; recombinant factor VIII

SUMMARY:
This trial is conducted in Japan. The aim of this clinical trial is to investigate the pharmacokinetics (the effect of the investigated drug on the body) and safety of turoctocog alfa (recombinant factor VIII (N8)) in Japanese subjects with haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects who have completed NN7008-3543
* No detectable inhibitors to factor VIII

Exclusion Criteria:

* Congenital or acquired coagulation disorders other than haemophilia A
* Planned surgery during the trial period
* Receipt of any investigational drug other than recombinant factor VIII (N8) within 30 days of trial product administration

Ages: 12 Years to 66 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Area under the curve | Infusion, 30 minutes
Incremental recovery | Infusion, 30 minutes
In vivo t1/2 | Infusion, 30 minutes
Total clearance (CL) | Infusion, 30 minutes

SECONDARY OUTCOMES:
Maximal concentration | at 15 minutes
Area under the curve | from time zero to last
Number of adverse events | from day -1 to day 3 (end of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (6):
- Japan (6):
  - Novo Nordisk Investigational Site, Itabashi-ku, Tokyo
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Maebashi-shi, Gunma
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Shizuoka-shi, Shizuoka
  - Novo Nordisk Investigational Site, Suginami-ku, Tokyo

REFERENCES:
- [Result] Jimenez-Yuste V, Lejniece S, Klamroth R, Suzuki T, Santagostino E, Karim FA, Saugstrup T, Moss J. The pharmacokinetics of a B-domain truncated recombinant factor VIII, turoctocog alfa (NovoEight(R)), in patients with hemophilia A. J Thromb Haemost. 2015 Mar;13(3):370-9. doi: 10.1111/jth.12816. Epub 2015 Feb 13. PMID 25495795
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com